CLINICAL TRIAL: NCT02912117
Title: Determining the Etiologic Diagnosis in Febrile Neutropenia Using the Karius Sequencing-based Infectious Disease Diagnostic Assay
Brief Title: Determining the Etiology of Febrile Neutropenia Using the Karius Sequencing-based Infectious Disease Diagnostic Assay
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 004-CL-01
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-03

CONDITIONS: Infection; Neutropenia
MeSH Terms: conditions — Infections; Neutropenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, observational study at Stanford University Hospital comparing the Karius Infectious Disease Diagnostic Sequencing Assay to the Final Microbiologic Diagnosis in Patients with Fever and Neutropenia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Are or will be admitted to Stanford University Hospital for fever and neutropenia
* Neutropenia - an absolute neutrophil count of <500 per cubic mm
* Documented fever or report of fever ≥38.3 or ≥38.0 on two episodes separated by at least one hour, resulting in hospitalization for febrile neutropenia

Exclusion Criteria:

* Inability to understand instructions and comply with study-related procedures
* Any condition that in the opinion of the treating physician will prevent the subject from completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted for fever and neutropenia at the Stanford University Hospital or patients who are admitted for chemotherapy who develop fever and neutropenia at Stanford University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value of the Karius Infectious Disease Diagnostic Sequencing Assay compared with standard clinical diagnosis | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley C Deresinski, MD, Principal Investigator — Stanford University; Jose G Montoya, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benamu E, Gajurel K, Anderson JN, Lieb T, Gomez CA, Seng H, Aquino R, Hollemon D, Hong DK, Blauwkamp TA, Kertesz M, Blair L, Bollyky PL, Medeiros BC, Coutre S, Zompi S, Montoya JG, Deresinski S. Plasma Microbial Cell-free DNA Next-generation Sequencing in the Diagnosis and Management of Febrile Neutropenia. Clin Infect Dis. 2022 May 3;74(9):1659-1668. doi: 10.1093/cid/ciab324. PMID 33870413